CLINICAL TRIAL: NCT02247726
Title: A Phase II Randomized, Observer-Blind, Placebo-Controlled, Study to Evaluate the Safety and Immunogenicity of a Respiratory Syncytial Virus (RSV) F Nanoparticle Vaccine With Aluminum, in Healthy Third-trimester Pregnant Women and to Assess the Impact of Maternal Immunization on Infant Safety Through One Year of Life
Brief Title: RSV F Vaccine Maternal Immunization Study in Healthy Third-trimester Pregnant Women.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RSV-M-203
Record Dates: First submitted 2014-09-16; First posted 2014-09-25 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV; Third Trimester; Maternal Immunization
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Group A (Placebo Comparator): Saline Placebo (0.5mL injection)
  Interventions: Drug: Saline Placebo (0.5mL injection)
- Treatment Group B (Experimental): RSV F vaccine with adjuvant (0.5mL injection)
  Interventions: Drug: RSV F vaccine (0.5mL injection)

INTERVENTIONS:
Drug: Saline Placebo (0.5mL injection)
  Other Names: 0.9% Sodium Choloride
  Arms: Treatment Group A
Drug: RSV F vaccine (0.5mL injection)
  Other Names: RSV F Protein with Aluminum adjuvant
  Arms: Treatment Group B

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of an RSV-F protein nanoparticle vaccine, with aluminum, in healthy third-trimester pregnant women and to assess the impact of maternal immunization on infant safety through one year of life.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women must meet all of the following criteria to be eligible to participate:

1. ≥18 and ≤40 years-of-age.
2. Singleton pregnancy of 33 to 35 weeks gestation on the day of planned vaccination.
3. Good general maternal health as demonstrated by:

   * Medical history (including history of adverse reactions to prior vaccines and allergies).
   * Physical examination including at least vital signs (blood pressure, pulse, respirations, and oral temperature); weight; height; examination of the HEENT, cardiovascular, pulmonary, gastrointestinal (abdominal), musculoskeletal, lymphatic, and dermatologic organ systems; and documentation of fetal heart tones.
   * Clinical laboratory parameters including normal blood urea nitrogen, creatinine, ALT, AST, total bilirubin, alkaline phosphatase (ALP), hemoglobin, white blood count, and platelet count; and serologic exclusion of infection with hepatitis B (HBV) and C (HCV) viruses and HIV (as required). Note that normal ranges for vital signs and clinical laboratory parameters will be based on third trimester values published in Sheffield et al. [2013] and/or reference ranges for the third trimester of pregnancy of the central laboratory.
4. Documentation that fulfills one of the following:

   * Detailed (level II) second trimester or later anatomic ultrasound with no significant anatomic or growth abnormalities identified; OR
   * Routine second trimester or later ultrasound with no significant anatomic or growth abnormalities identified, PLUS at least one of the following:

     * Normal first trimester screening (based on ultrasound + serum analytes); or
     * Normal cell-free fetal DNA; or
     * Normal chorionic villus sampling (CVS) or amniocentesis; or
     * Normal second trimester maternal serum quadruple screen; or
     * Normal first and second trimester screening using integrated, sequential, or contingency approach; or
     * Abnormal first or second trimester screening followed by normal CVS, amniocentesis, or cell-free fetal DNA.
5. Able to understand, and both willing and physically able to comply with study procedures. This includes anticipation of reasonable geographic proximity to the study clinic and adequate transportation to comply with scheduled and unscheduled study follow-up visits.
6. Able and willing to provide written informed consent for themselves and infant.

Exclusion Criteria:

Pregnant women will be excluded if there is historical, physical examination, or laboratory evidence of any of the following criteria:

1. Symptomatic cardiac or pulmonary disease requiring chronic drug therapy, including hypertension and asthma. Asthma will be exclusionary if the subject is receiving chronic systemic glucocorticoids at any dose or inhaled glucocorticoids at any dose >500µg per day of beclamethasone or fluticasone, or >800μg per day of budesonide.
2. Pre-pregnancy body mass index (BMI) of ≥35 or <18.5.
3. Hemoglobinopathy (including known sickle trait or thalassemias, even if asymptomatic) or blood dyscrasias.
4. Hepatic or renal dysfunction.
5. Established diagnosis of seizure disorder, regardless of therapy.
6. Auto-immune disease or known immunodeficiency syndrome.
7. Endocrine disorders, including (but not limited to) hyperthyroidism, untreated hypothyroidism, and glucose intolerance (e.g., diabetes mellitus type 1 or 2) antedating pregnancy, or occurring during pregnancy and requiring interventions other than diet for control.
8. History of major gynecologic or major abdominal surgery, including bariatric surgery.
9. Known HIV, HBV, or HCV infection, as assessed by serologic tests conducted during the current pregnancy or as a procedure during the screening period of the study.
10. Primary genital herpes simplex (HSV) infection during the current pregnancy.
11. Current alcohol or drug abuse.
12. Documentation that current pregnancy results from fertility treatments, rape, or incest.
13. Documentation that the infant will be a ward of the state or be released for adoption.
14. Neuro-psychiatric illness deemed likely to interfere with protocol compliance, safety reporting, or receipt of pre-natal care; or requiring treatment with psychotropic drugs.
15. History/presence of deep venous thrombosis or thromboembolism, or the use of anticoagulants during pregnancy.
16. Untreated red blood cell allo-immunization.
17. Prior stillbirth or neonatal death, or multiple (≥3) spontaneous abortions.
18. Prior preterm delivery ≤34 weeks gestation or having ongoing intervention (medical/surgical) in current pregnancy to prevent preterm birth.
19. Greater than five (5) prior deliveries.
20. Previous infant with a known genetic disorder or major congenital anomaly.
21. Receipt of investigational drugs or immune globulins (with the exception of prophylactic anti-Rho D immune globulin) within six (6) months prior to the administration of the study vaccine.
22. Chronic administration (defined as more than 14 continuous days) of immunosuppressants or other immune-modifying drugs within 6 months prior to the administration of the study vaccine. An immunosuppressant dose of glucocorticoid will be defined as a systemic dose ≥10mg of prednisone per day or equivalent. The use of topical, inhaled, and nasal glucocorticoids will be permitted except for the limit established in exclusion criterion #1.
23. Any other physical, psychiatric or social condition which may, in the investigator's opinion, increase the risks of study participation to the maternal subject or the fetus/infant; or may lead to the collection of incomplete or inaccurate safety data.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Counts and percentage of subjects with solicited injection site and systemic reactogenicity within seven days of vaccination. | Day 0 to Day D+180
  In Maternal Subjects
Counts and percentage of subjects with unsolicited (local and systemic) adverse events (AE), unscheduled medically-attended adverse events (MAEs), and serious adverse events (SAEs) through delivery and six (6) months thereafter. | Day 0 to Day D+180
  In Maternal Subjects
Clinical safety laboratory assessments of select serum chemistry and hematology parameters through delivery. | Screening to Day 14
  In Maternal Subjects
Counts and percentage of subjects with post-immunization onset of specific complications of third-trimester pregnancy and delivery | Day 0 to Day 28 - 42
  In Maternal Subjects
Counts and percentage of term healthy infants appropriate for gestational age. | Day 28 - 42
  In Infant subjects
Neonatal SAEs (including congenital anomalies, respiratory failure, fever/infection, and neonatal death or other adverse events/complications that necessitate extended hospitalization). | Birth to Day 365
  In Infant Subjects
Growth and development over one year | Birth to Day Day 365
  In Infant Subjects
Counts and proportion of infants with unsolicited adverse events | Birth to Day 365
  In Infant Subjects
Counts and proportions of infants with medically-attended RSV lower respiratory tract infection (LRTI), and age of onset of those infections. | Birth to Day 365
  In Infant Subjects

SECONDARY OUTCOMES:
Immunogenicity as assessed by serum IgG antibody titers specific fro the F-Protein antigen. | Birth to Day 180
  In Infant Subjects
Serum antibody titers inhibiting binding of labeled palivizumab to RSV F protein. | Birth to Day 180
  In Infant Subjects
Serum microneutralization (MN) titers against RSV/A and B.previously referenced, but based on GMT. | Birth to Day 180
  In Infant Subjects

OTHER OUTCOMES:
Counts and proportions of maternal subjects with RSV-related respiratory illness as detected by active and passive surveillance. | Day 0 to Day 180
  In Maternal Subjects
Counts and proportions of infants with non-medically attended RSV-related respiratory illness as detected by active and passive surveillance. | Birth to Day 365
  In Infant Subjects
Counts and proportions of infants with medically attended, non-RSV LRTI as assessed by multiplex real time (RT)-PCR. | Birth to Day 365
  In Infant Subjects

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (7):
- United States (7):
  - Advanced Specialty Research, Nampa, Idaho
  - Hutchinson Clinic, P.A., Hutchinson, Kansas
  - University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Meridian Clinical Research, Norfolk, Nebraska
  - Duke University, Durham, North Carolina
  - Magee- Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Munoz FM, Swamy GK, Hickman SP, Agrawal S, Piedra PA, Glenn GM, Patel N, August AM, Cho I, Fries L. Safety and Immunogenicity of a Respiratory Syncytial Virus Fusion (F) Protein Nanoparticle Vaccine in Healthy Third-Trimester Pregnant Women and Their Infants. J Infect Dis. 2019 Oct 22;220(11):1802-1815. doi: 10.1093/infdis/jiz390. PMID 31402384
- See also: Novavax, Inc. — http://novavax.com